CLINICAL TRIAL: NCT07121192
Title: A Phase 2a Randomized, Observer-Blind, Study to Evaluate the Immunogenicity and Safety of mRNA-Based Multivalent Seasonal Influenza Vaccine Candidates in Adults 18 Years of Age And Older
Brief Title: A Study to Assess the Immune Response and Safety of a Vaccine Against Influenza in Adults 18 Years of Age and Older
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 300356; 2025-522278-35 (EudraCT Number)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Influenza, Human
Keywords: Influenza; Human; Virus Diseases; Infections; mRNA vaccine; Younger Adults; Older Adults; multivalent seasonal influenza vaccine
MeSH Terms: conditions — Influenza, Human; Virus Diseases; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an Observer-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Flu mRNA_1_YA (Experimental): Eligible Younger Adults (YA) participants receive a single dose of Flu mRNA Formulation A (GSK6479720A) as study intervention at Day 1.
  Interventions: Biological: Flu mRNA (Formulation A)
- Flu mRNA_2_YA (Experimental): Eligible YA participants receive a single dose of Flu mRNA Formulation B (GSK6479715A) as study intervention at Day 1.
  Interventions: Biological: Flu mRNA (Formulation B)
- Comparator_1_YA (Active Comparator): Eligible YA participants receive a single dose of comparator 1 at Day 1.
  Interventions: Combination Product: Comparator 1
- Comparator_2_YA (Active Comparator): Eligible YA participants receive a single dose of comparator 2 at Day 1.
  Interventions: Combination Product: Comparator 2
- Flu mRNA_1_OA (Experimental): Eligible Older Adults (OA) participants receive a single dose of Flu mRNA Formulation A (GSK6479720A) as study intervention at Day 1.
  Interventions: Biological: Flu mRNA (Formulation A)
- Flu mRNA_2_OA (Experimental): Eligible OA participants receive a single dose of Flu mRNA Formulation B (GSK6479715A) as study intervention at Day 1.
  Interventions: Biological: Flu mRNA (Formulation B)
- Comparator_1_OA (Experimental): Eligible OA participants receive a single dose of comparator 1 at Day 1.
  Interventions: Combination Product: Comparator 1
- Comparator_2_OA (Active Comparator): Eligible OA participants receive a single dose of comparator 2 at Day 1.
  Interventions: Combination Product: Comparator 2
- Comparator_3_OA (Active Comparator): Eligible OA participants receive a single dose of comparator 3 at Day 1.
  Interventions: Combination Product: Comparator 3

INTERVENTIONS:
Biological: Flu mRNA (Formulation A) — One dose of Flu mRNA (Formulation A) received intramuscularly.
  Other Names: GSK6479720A
  Arms: Flu mRNA_1_OA; Flu mRNA_1_YA
Biological: Flu mRNA (Formulation B) — One dose of Flu mRNA (Formulation B) received intramuscularly.
  Other Names: GSK6479715A
  Arms: Flu mRNA_2_OA; Flu mRNA_2_YA
Combination Product: Comparator 1 — One dose of Comparator 1 received intramuscularly.
  Arms: Comparator_1_OA; Comparator_1_YA
Combination Product: Comparator 2 — One dose of Comparator 2 received intramuscularly.
  Other Names: Click here to enter text.
  Arms: Comparator_2_OA; Comparator_2_YA
Combination Product: Comparator 3 — One dose of Comparator 3 received intramuscularly.
  Arms: Comparator_3_OA

SUMMARY:
"The purpose of this study is to assess the reactogenicity, safety and immune response of GlaxoSmithKlines (GSK) messenger RNA (mRNA)-based multivalent seasonal influenza vaccine candidates administered in healthy younger and older adults."

ELIGIBILITY:
Inclusion Criteria:

1. Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiary, attendance to study contacts and study site visits, and ability to access and utilize a phone or other electronic communications) independently or with the assistance of a caregiver.
2. Written (physically, or digitally) informed consent obtained from the participant prior to performance of any study-specific procedure.
3. A male or female at least 18 YOA at the time of the screening.
4. Healthy participants or medically stable patients as established by medical history, and clinical examination. Participants with chronic medical conditions with or without specific treatment (e.g., chronic metabolic, cardiac, pulmonary, renal, neurologic, and hematologic diseases) are allowed to participate in this study, if considered by the investigator as medically stable. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during 3 months before enrollment.
5. Female participants of non-childbearing potential may be enrolled in the clinical study.
6. Female participants of childbearing potential may be enrolled in the clinical study, if the participant:

   * Has practiced adequate contraception for at least 4 weeks prior to the study intervention administration, and
   * Has a negative urine pregnancy test within 24 hours prior to the study intervention administration, and
   * Has agreed to continue adequate contraception for at least 8 weeks after study intervention administration.
7. Body mass index (BMI) between18 kg/m^² and 33kg/m^².

Exclusion Criteria:

1. Where applicable, FDA toxicity grades will be exclusionary.
2. Immunosuppressive or immunodeficient conditions by history/exam; stable HIV-positive individuals on therapy can participate.
3. History of Guillain-Barré Syndrome within 6 weeks of receiving any vaccine.
4. Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study (e.g., life-threatening disease likely to limit survival to less than 1 year).
5. Hypersensitivity to latex.
6. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
7. History of hypersensitivity or severe allergic reaction to any previous influenza vaccine.
8. History of hypersensitivity or severe allergic reaction to any previous mRNA vaccine.
9. History of or current suspicion of myocarditis or pericarditis, or medical issues increasing such risks.
10. Condition that in the judgment of the investigator would make intramuscular injection unsafe.
11. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the clinical study.
12. History of confirmed influenza infection by local health authority-approved testing methods within 180 days prior to study intervention administration.
13. Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study intervention(s) during the period beginning 28 days before the dose of study intervention(s) (Day -28 to Day 1), or their planned use during the study period.
14. Administration of an influenza vaccine within 180 days before the study intervention administration or planned administration prior to Visit 4 (Day 29) during the study.
15. Administration of any non-live attenuated non-study vaccine in the period starting 14 days before the study intervention administration, or planned administration within 14 days after study intervention administration.
16. Administration of any live attenuated and/or mRNA non-study non-influenza vaccine in the period starting 28 days before the study intervention administration, or planned administration within 28 days after study intervention administration.
17. Chronic administration of immune-modifying drugs.
18. Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the study intervention, or planned administration during the study period.
19. Administration of anti-tumoral medication during the period starting 90 days before the study intervention or planned administration during the study period.
20. Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention.
21. Any study personnel or their immediate dependents, family, or household members.
22. Has a history of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
23. Participant is pregnant.
24. Participant is breastfeeding or will (re)start breastfeeding during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) Ratio of Antigen 1 Titer | At Day 29
Geometric Mean Increase (GMI) of Antigen 1 Titer | From Day 1 to Day 29
Percentage of Participants with Antigen 1 Seroconversion Rate (SCR) | From Day 1 to Day 29
Percentage of Participants with Antigen 1 Seroprotection Rate (SPR) | At Day 1 and Day 29
Number of Participants with Solicited Administration Site Adverse Events (Aes) | From Day 1 to Day 7
  The solicited administration site AEs considered are pain, redness, swelling and lymphadenopathy.
Number of Participants with Solicited Systemic Aes | From Day 1 to Day 7
  The solicited systemic AEs considered are fever, headache, fatigue, myalgia, arthralgia and chills. Fever is defined as temperature greater than or equal to (>=) 38 °C/100.4°F regardless the location of measurement.
Number of Participants with Unsolicited Aes | From Day 1 to Day 28
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Number of Participants with Serious Adverse Events (SAEs) | From Day 1 to Day 181 (study end)
  SAE is an AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or other situations that are considered serious per medical or scientific judgment.
Number of Participants with Adverse Events of Special Interest (AESIs) | From Day 1 to Day 181 (study end)
Number of Participants with Medically Attended Adverse Events (MAAEs) | From Day 1 to Day 181 (study end)
  A MAAE is an AE for which the participant received medical attention including any symptom or illness requiring hospitalization, or an emergency room visit, or visit to/by a healthcare professional.
Number of Participants with any Laboratory abnormalities | From Day 1 to Day 29
  Click here to enter text.

SECONDARY OUTCOMES:
GMT Ratio of Antigen 2 Titer | At Day 29
GMI of Antigen 2 Titer | From Day 1 to Day 29
Percentage of Participants with Antigen 2 SCR | From Day 1 to Day 29

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Fair Oaks, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Carson City, Nevada
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, North Charleston, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, DeSoto, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf